CLINICAL TRIAL: NCT01493635
Title: An International, Multicentre, Open Randomised Parallel Group Trial Comparing a Two Step Approach for Cancer Pain Relief With the Standard Three Step Approach of the WHO Analgesic Ladder in Patients With Cancer Pain Requiring Step 2 Analgesia.
Brief Title: Two Step Versus the Standard Three Step Approach of the WHO Analgesic Ladder for Cancer Pain Relief.
Acronym: TVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 11/SS/0079
Record Dates: First submitted 2011-12-15; First posted 2011-12-16 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2015-12

CONDITIONS: Cancer; Pain
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard 3 Step approach. (Active Comparator): Standard 3 Step approach of the WHO analgesic ladder (Step 1 - Step 2 - Step 3).
  Interventions: Other: analgesic ladder
- 2 Step approach. (Experimental): 2 Step approach of the WHO analgesic ladder (Step 1 - Step 3).
  Interventions: Other: analgesic ladder

INTERVENTIONS:
Other: analgesic ladder — Patients will be managed according to the standard 3 Step approach of the WHO analgesic ladder (Step 1 - Step 2 - Step 3).
  Arms: Standard 3 Step approach.
Other: analgesic ladder — Patients managed according to the WHO analgesic ladder bypassing Step 2, i.e. patients will move from Step 1 of the WHO analgesic ladder to Step 3.
  Arms: 2 Step approach.

SUMMARY:
The World Health Organization analgesic ladder for cancer pain relief is an internationally used approach to managing cancer pain. Patients generally start on Step 1 of the ladder (paracetamol). As pain increases or is not well controlled on this, they progress to Step 2 which involves a stronger pain killer (weak opioid such as codeine). If pain is still not controlled they progress to Step 3 of the ladder which is a strong opioid (such as morphine). Work to date has suggested that Step 2 may be unnecessary and most patients usually require Step 3 analgesia. The TVT trial aims to examine the standard approach (Step 1-Step2-Step-3) versus a two step approach (Step 1-Step 3).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and over.
* Patient has a cancer diagnosis (based on radiological, histological, cytological, or operative evidence). Those with haematological malignancies are eligible.
* Cancer related pain - which in the opinion of the clinician is caused by the presence of tumour or metastases.
* Average pain score > 4, on a numerical rating scale from 0-10, requiring step 2 analgesia (weak opioid).
* Patient is able to comply with trial procedures.

Exclusion Criteria:

* Patients who have received radiotherapy in the previous 6 weeks or are planned to receive radiotherapy during the trial period where in either case, it is expected to affect pain during the trial period.
* Pain due to surgery in the preceding 4 weeks.
* Life expectancy less than two months (based on clinical impression).
* Patients with psychotic disorders or cognitive impairment.
* Patients who have received regular doses (scheduled doses - NOT as required dosing) of weak or strong opioids in the preceding two weeks.
* Patients using immediate release opioids > 2 doses/24 hours, in the previous 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2012-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Time to achieving stable pain control, where stable pain control is defined as the first day of three consecutive days with average pain score less than or equal to 3 using scores from the Patient Diary and patient assessments. | Up to 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Marie Fallon, Principal Investigator — University of Edinburgh
Locations (1):
- Western General Hospital, Edinburgh, United Kingdom